CLINICAL TRIAL: NCT03583112
Title: Investigation of the Changes of Brain Structure and Function in Premature Ejaculation Patients and the Effects of Dapoxetine on Central Neural Activity in Premature Ejaculation Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xidian University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 81471811
Record Dates: First submitted 2018-05-30; First posted 2018-07-11 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2018-05

CONDITIONS: Premature Ejaculation
MeSH Terms: conditions — Premature Ejaculation | interventions — dapoxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapoxetine (Active Comparator): In this group, patients received one dapoxetine hydrochloride tablet before MRI scan.
  Interventions: Drug: Dapoxetine Hydrochloride Tablet
- Placebo (Placebo Comparator): In this group, patients received placebo tablet before MRI scan.
  Interventions: Drug: Placebo Tablet

INTERVENTIONS:
Drug: Dapoxetine Hydrochloride Tablet — oral one dapoxetine hydrochloride tablet before MRI scan
  Arms: Dapoxetine
Drug: Placebo Tablet — oral one placebo tablet before MRI scan.
  Arms: Placebo

SUMMARY:
Lifelong premature ejaculation (LPE) is a common male sexual dysfunction with a high prevalence in global. Up to now, the etiology of LPE remains unclear. In recent years, dapoxetine, a highly potent serotonin-transporter inhibitor, has been used for treating premature ejaculation. However, the underlying mechanism of dapoxetine was unknown. Recently, with widespread use of neuroimaging techniques, like positron emission tomography and magnetic resonance imaging (MRI) in basic science, researchers can acquire human data on cerebral base of human sexual behavior, not only in normal subjects but also in patients with sexual dysfunction. Therefore, in order to further understand the biological mechanism of LPE and the brain targets of dapoxetine, the present study would investigate the brain changes of LPE and the effect of dapoxetine on brain activation by using MRI technology.

ELIGIBILITY:
Inclusion Criteria:

* right-handed male Chinese volunteers
* intravaginal ejaculatory latency time within 1 min
* premature ejaculation diagnostic tool score >11 for patients, but <5 for each control.
* patients who never received dapoxetine hydrochloride or other SSRI drugs

Exclusion Criteria:

* smokers
* had medical，neurological or psychiatric disorders
* had alcohol, nicotine, or drug abuse
* received any treatment at least 2 weeks before the experiment

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-07-10 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Resting-state brain function measured by Functional magnetic resonance imaging | One day
  We will use several indicators to assess the resting-state brain function based on fMRI analysis, including regional homogeneity,Amplitude of Low Frequency Fluctuations, and functional connectivity.

CONTACTS AND LOCATIONS:
Overall Officials: Gao, Principal Investigator — The ART Center, The Northwest Women's and Children's Hospital
Locations (1):
- The ART Center, The Northwest Women's and Children's Hospital,, Xi'an, Shaanxi, China